CLINICAL TRIAL: NCT06409468
Title: Safety and Efficacy of NovoMatrix in Gingival Recession Coverage /A Pilot Clinical and Histological Case Series/
Brief Title: NovoMatrix in Gingival Recession Coverage: Case Series
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Novomatrix
Record Dates: First submitted 2024-05-09; First posted 2024-05-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronally Advanced Tunnel with NovoMatrix (Experimental): Gingival Augmentation Procedure using NovoMatrix + Coronally Advanced Tunnel
  Interventions: Procedure: Subperiostal tunnel in conjunction with Novomatrix

INTERVENTIONS:
Procedure: Subperiostal tunnel in conjunction with Novomatrix — An intrasulcular incision on the tooth with recession and on each adjacent tooth. Subperiosteal pouches dissected apically for about 6-8 mm facial to the 3 teeth and connected by extension of the subperiosteal dissection into the interdental areas to create a tunnel. NovoMatrix trimmed to a vertical dimension of 7-8 mm and a horizontal length to completely over the exposed roots and extend laterally to the root line angles of the adjacent teeth. The graft inserted into the tunnel and aligned. Both the overlying tissue and graft positioned 1mm coronally to the level of the cementoenamel junction and secured with a 6-0 resorbable sling suture.

SUMMARY:
Twenty patients seeking treatment for gingival recession coverage, ranging from 20-70 years of age with multiple Miller Class I or II buccal gingival recessions (depth≥3 mm, at least 3 adjacent teeth) will be recruited for this study. Five patients within the study patient pool looking for further orthodontic or restorative treatment that requires removal of one single rooted tooth within the study site of interest will be selected for histological sample removal. All procedures performed in this study will be executed according to established routine protocols, with the exception of block biopsies of one hopeless tooth per patient (total of 5 patients) at 6 months.

DETAILED DESCRIPTION:
Patient Selection Ten patients requiring gingival recession coverage (Miller Class I or II with multiple buccal gingival recession ≥3 mm, at least 3 adjacent teeth) will be enrolled and prepared for surgery in accordance with accepted dental practice guidelines (including informed consent). The appropriate demographic and medical history, physical examination and radiographs will be performed and recorded. Other therapies will not be withheld from the patient if the investigator determines that they are appropriate. Any adverse events will be recorded and reported on the appropriate case report form. Any and all complications will be addressed in an appropriate manner at the discretion of the investigator.

Inclusion Criteria

1. Male or female, between 20-70 years of age, who request gingival augmentation or recession coverage.
2. Subjects who are willing to sign an informed consent, participate and return for follow-up visits.
3. Subjects without significant medical history and currently not on medications that might complicate treatment outcomes.
4. Subjects demonstrating good oral hygiene (FMPS, FMBS less than 20%).

Exclusion Criteria

1. Subjects who do not meet all the inclusion criteria or who will not cooperate with the protocol schedule.
2. Subjects who received and failed a previously placed autogenous graft.
3. Subjects who have significant untreated periodontal disease, caries, infection or chronic inflammation in the oral cavity within two adjacent tooth positions of the clinical trial area.
4. Subjects who have used nicotine-containing products within 3 weeks prior to surgery.
5. Subjects who are insulin-dependent diabetic or if their Hgb1c levels > 6.5%.
6. Subjects who have had a history of malignancy within the past 5 years (except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma).
7. Subjects who are nursing or pregnant.
8. Subjects who are presently taking medications (except estrogen/progesterone therapy) or those who are undergoing treatment that in known to have an effect on bone turnover.
9. Subjects who have diseases that affect bone metabolism (excluding idiopathic osteoporosis).
10. Subjects with a history of an autoimmune disease, documented allergy or multiple allergies to any component of the agents used in this study.
11. Acutely infected mucogingival defect site.

Gingival Augmentation Procedure All surgical procedures will be performed on an outpatient basis. A full periodontal and radiographic examination (periapical radiographs) will be conducted for each patient presurgically. Before surgery, subjects will receive professional dental cleaning. At the time of surgery, local anesthesia will be administered and the surgical procedure (estimated to require approximately two hours) will be performed.

Immediately prior to and 1, 3, 6 months after surgery, the following measurements will be made using a periodontal probe (UNC-15) at the facial aspect of each tooth along the mucogingival defect extension: plaque index (PI), gingival index (GI), probing depth (PD), recession depth (RD), recession width (RW) and keratinized tissue width (KW). Keratinized tissue thickness (KT) will be measured directly using sterile Kerr-files, as well as indirectly by means of an ultrasonic device (PIROP Biometric scanner G-scan, Echoson, Poland). Intraoral scanning will be performed to assess surface changes (Emerald, Planmeca, Finland). Resistance to muscle pull (based on whether the free gingival margin of the tissue facial to the site moved when the adjacent cheek was retracted) will be evaluated. Pre- and postoperative blood flow will be assessed using a Laser Speckle Contrast Imaging device (785nm PeriCam PSI HR System, Perimed AB, Sweden) at Day 0, 1, 4, 7, 10, 14, Month 1, 3, 6. Any adverse events such as local or systemic reactions will be recorded. After giving both verbal and written post-surgical instructions to the patient, the investigator will release the patient when it is medically appropriate.

Pre- and post-surgical clinical examinations will be performed, and oral hygiene instructions reinforced at each post-surgical visit. Following surgery the patients will be seen at Day 0, 1, 4, 7, 10, 14, Month 1, 3, 6 until biopsy at 6 month post surgery (periapical radiographs will be taken at baseline and at 6 month).

Block biopsy removal After a healing period of 6 months, a block biopsy will be harvested under local anesthesia from each patient and immediately immersed in a fixative solution (estimated to require approximately two hours). The biopsied sites will be repaired with both hard and soft tissue grafting as necessary. The duration of the proposed study from treatment (gingival augmentation procedure) to biopsy is up to 6 months.

Implant placement 9 months after biopsy removal implant placement will be carried out in local anesthesia following mucoperiosteal flap elevation. Alternatively, orthodontic gap closure or conventional prosthetic reconstruction can be performed depending on individual needs.

Efficacy Evaluations

Soft Tissue Evaluation Plaque index (PI), gingival index (GI), probing depth (PD), recession depth (RD), recession width (RW) and keratinized tissue width (KW) will be recorded immediately prior to and 1, 3, 6 months after surgery. In 5 patients, a block biopsy of treated tooth will be collected and analyzed.

Pre-Surgical Phase Necessary diagnostic information will be gathered (Clinical photographs, periapical radiographs and etc.).

Surgical Phase Initial periodontal therapy including oral hygiene instruction and adult prophylaxis will be performed before the surgery. The surgery will not be performed until satisfactory plaque control is achieved. The patients will take Amoxicillin 1000mg 1 hour before surgery, then 2x1000mg daily for the next 7 days. The tooth scheduled for extraction for either orthodontic or restorative reason will be anesthetized with local anesthesia (Ultracain DS Forte, Sanofi Aventis, France). Immediately after local anesthesia, root debridement with hand instruments and removal of the smear layer with an EDTA solution will be performed. An intrasulcular incision will be made on the tooth with recession and on each adjacent tooth. Subperiosteal pouches will be dissected apically for about 6-8 mm facial to the 3 teeth and connected by extension of the subperiosteal dissection into the interdental areas to create a tunnel. The papillae will be separated from the interdental bone crests by blunt dissection. The tunnel will be extended apically about 6-8 mm by sharp dissection immediately supraperiosteally flap to ensure the tension-free coronal displacement of the tunnel. NovoMatrix will be trimmed to a vertical dimension of 7-8 mm and a horizontal length to completely over the exposed roots and extend laterally to the root line angles of the adjacent teeth. The graft will be inserted into the tunnel and aligned so that the coronal border of the graft is level with the coronal border of the overlying tissue. Both the overlying tissue and graft will be positioned 1mm coronally to the level of the cementoenamel junction and secured with a 6-0 resorbable sling suture (Monolac, Chirmax, Czech Republic; resorption time 4 weeks). Similar surgical approaches will be rendered for the control group. Two weeks after surgery the grafted area will be carefully cleaned with 0,2% chlorhexidine solution (Curasept, Curaden, Sweden). The sutures will be removed at 4 weeks, if necessary. Patients will be seen at at Day 0, 1, 4, 7, 10, 14, Month 1, 3, 6 until biopsy at 6- month post surgery to monitor healing and plaque control.

Six months after gingival augmentation procedure, a block biopsy will be harvested under local anesthesia from each patient. The biopsy area will be reconstructed with both hard and soft tissue grafting as necessary.

Post-Surgical Care The patients will be instructed not to brush or floss the surgical site(s) until 2-3 weeks when the graft has become stabilized by healing. Patients will be instructed to rinse with chlorhexidine mouth rinse (0.2%) 2-3 times daily for 2-3 weeks. Any adverse effects will be recorded.

Management of Post-Surgical Oral Pain Post-surgical discomfort will be divided into mild, moderate and severe levels and requires a subjective assessment by the investigator based on his knowledge of the surgical procedure to be performed and the presenting signs and symptoms of the patient. Treatment of the source of pain is usually the best management. If infection is present, treatment of the infection will directly alleviate the patient's discomfort.

The following medications will be given to provide relief follows: 3x400mg Ibuprofen (Advil Ultra Forte, Pfizer, USA) during the first 2-3 days after surgery. All prescription pain medications will be closely monitored for efficacy, and dosages altered if the pain persists or requires a higher level formulation.

Follow-Up Evaluations Patients will be seen for post-operative evaluations at Day 0, 1, 4, 7, 10, 14, Month 1, 3, 6 until the biopsies are obtained. Localized supragingival scaling, polishing and oral hygiene reinforcement will be performed according to individual needs at each visit. At 3 and 6 months, periodontal maintenance will be performed which includes an evaluation of the dental plaque and the gingival condition for the whole mouth. Photographs of the treated sites will be obtained.

Biopsy All biopsies will be placed into fixative solution (which will be supplied), clearly labeled and sent via Express Mail or hand delivered to the histological lab. All results and corresponding documentation, including both histological and clinical findings and radiographs, should be sent by Express Mail to the histological lab, who will be responsible for compiling all data and preparation of the final study report.

Study Discontinuation

Participants will be removed from the study prematurely if:

* The subject requests to be withdrawn from the study.
* The principal investigator decides that it is in the subject's best interest.
* The subject is noncompliant with the protocol.

Adverse Events An adverse event is defined as any untoward medical occurrence in a clinical investigation treatment and does not necessarily have a causal relationship with this treatment. An adverse event can, therefore, be any unfavorable and unintended sign of symptom, or disease temporarily associated with the use of an investigational product, whether or not related to the investigational product. All patients will be prepared for surgery in accordance with accepted dental practice. The appropriate demographic and medical history, physical examination, diagnostic laboratory and radiographic work will be performed and recorded.

Confidentiality All information provided to the Principal Investigator by BioHorizons or their designates including non-clinical data, protocols, clinical research findings, and verbal and written information, will be kept strictly confidential and confined to the clinical personnel involved in conducting the study. It is recognized that this information may be related in confidence to the Ethics Committee. In addition, no reports or information about the study or its progress will be provided to anyone not involved in the study other than to BioHorizons or their designates (if required by law).

Ethical guidelines The study will be carried out in a single center (Department of Peridontology, Semmelweis University, Budapest, Hungary). Following screening, prior to surgery, written informed consents will be collected from participants. The study protocol and written informed consent will be approved by the Semmelweis University's Regional, Institutional Scientific and Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 20-70 years of age, who request gingival augmentation or recession coverage.
* Subjects who are willing to sign an informed consent, participate and return for follow-up visits.
* Subjects without significant medical history and currently not on medications that might complicate treatment outcomes.
* Subjects demonstrating good oral hygiene (FMPS, FMBS less than 20%).

Exclusion Criteria:

* Subjects who do not meet all the inclusion criteria or who will not cooperate with the protocol schedule.
* Subjects who received and failed a previously placed autogenous graft.
* Subjects who have significant untreated periodontal disease, caries, infection or chronic inflammation in the oral cavity within two adjacent tooth positions of the clinical trial area.
* Subjects who have used nicotine-containing products within 3 weeks prior to surgery.
* Subjects who are insulin-dependent diabetic or if their Hgb1c levels > 6.5%.
* Subjects who have had a history of malignancy within the past 5 years (except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma).
* Subjects who are nursing or pregnant.
* Subjects who are presently taking medications (except estrogen/progesterone therapy) or those who are undergoing treatment that in known to have an effect on bone turnover.
* Subjects who have diseases that affect bone metabolism (excluding idiopathic osteoporosis).
* Subjects with a history of an autoimmune disease, documented allergy or multiple allergies to any component of the agents used in this study.
* Acutely infected mucogingival defect site.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Histology | 6 months
  histologically evaluate the quality of newly formed soft tissues 6 months following gingival recession coverage utilizing NovoMatrix.

SECONDARY OUTCOMES:
Postoperative Blood Perfusion changes | Day 0, 1, 4, 7, 10, 14, Month 1, 3, 6
  Measurements are done by Laser Speckle Contrast Imaging system. Measurements are done at different timepoints. Region of Interests (ROI) are selected and created in PimSoft, the systems own software, which gives a number, called Perfusion Unit, that correlates with the superficial red blood cell movements.
Recession depth | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe, at the midbuccal surface in mm.
Recession width | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe, at the midbuccal at the line of CEJ in mm.
Papilla-Contact point distance | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe in mm.
Papilla width | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe in mm at the line of the CEJ.
Probing Pocket Depth | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe in mm at 3 surfaces, Distal, Midbuccal and Mesial.
Width of the Keratinized tissue (KTW) | Baseline, 1, 3, 6 months and 1 year
  Measured by UNC-15 probe in mm at 3 surfaces, Distal, Midbuccal and Mesial.
Volumetric changes | Baseline, 1, 3, 6 months and 1 year
  Measured in mm. Intraoral scanning is performed to assess volumetric changes (Emerald, Planmeca, Finland). Data is collected in an STL file, and later evaluated by superimposition.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Windisch, Profesor, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Faculty of Dentistry, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No